CLINICAL TRIAL: NCT00117364
Title: Effect of SACCHACHITIN on Healing of Chronic Wound ---A Clinical Trial
Brief Title: Effect of SACCHACHITIN on Healing of a Chronic Wound
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EIRB NO 940318-3
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2005-07-06 (Estimated); Status verified 2005-06

CONDITIONS: Wounds
Keywords: chronic ulcer; poor healing; The patients with a poorly healed wound, in which skin graft is clinically indicated, are included in this study
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Drug: SACCHACHITIN patch

SUMMARY:
SACCHACHITIN gel, prepared from the waste residue of the fruiting body of Ganoderma tsugae, was used in a previous study to enhance skin wound healing in animal models. In the present study, the effects of the gel on the activity of matrix metalloproteinases (MMPs) and vascular endothelial growth factor (VEGF) as well as on the healing of skin wounds in humans are estimated by a clinical trial.

The hypothesis regarding the poor healing of the wound is the over-expression of MMP and the inhibition of the angiogenic factors. From the previous animal study, the effect of SACCHACHITIN was to inhibit the activity of MMP and stimulation of VEGF and we try to prove the effect over the human wounds from this clinical trial.

Patients with a poorly healed wound, in which skin graft is clinically indicated, are included in this study. The exudates from the wound are collected and analyzed for the activity and concentration of VEGF and MMP. The change of the healing process is recorded.

Positive results are expected from the clinical trial and the patients will get another choice for the treatment of the chronic wound other than skin grafting.

DETAILED DESCRIPTION:
SACCHACHITIN gel, prepared from the waste residue of the fruiting body of Ganoderma tsugae, was used in a previous study to enhance skin wound healing in animal models. In the present study, the effects of the gel on the activity of matrix metalloproteinases (MMPs) and vascular endothelial growth factor (VEGF) as well as on the healing of skin wounds in humans are estimated by a clinical trial.

The hypothesis regarding the poor healing of the wound is the over-expression of MMP and the inhibition of the angiogenic factors. From the previous animal study, the effect of SACCHACHITIN was to inhibit the activity of MMP and stimulation of VEGF and we try to prove the effect over the human wounds from this clinical trial.

Patients with a poorly healed wound, in which skin graft is clinically indicated, are included in this study. The exudates from the wound are collected and analyzed for the activity and concentration of VEGF and MMP. The change of the healing process is recorded.

Positive results are expected from the clinical trial and the patients will get another choice for the treatment of the chronic wound other than skin grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a poorly healed wound, in which skin graft is clinically indicated

Exclusion Criteria:

* Skin infection
* Vital signs unstable

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Bin Chen, MD, Principal Investigator — Min-Sheng General Hospital
Locations (1):
- Min-Sheng General Hospital, Taoyuan, Taiwan